CLINICAL TRIAL: NCT04265976
Title: Emergency Departement (ED) Hypernatremia. Prognostic Factors and Epidemiology. About a Single-center Prospective Study
Brief Title: ED Hypernatremia. Prognostic Factors and Epidemiology.
Acronym: NATSAU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2019/448
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Hypernatremia
MeSH Terms: conditions — Hypernatremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluate the 1-month mortality of patients who proceed a blood sample while in the ED with an hypernatremia (>145 mmol/l). This prospective study will try to show several prognostic factors, and show the epidemiology of hypernatremia in this single center evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Natremia > 145 mmol/l

Exclusion Criteria:

* Age < 18 years
* Refusal

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Every >18 years old patient from who a blood sample was taken in the ED with a natremia > 145 mmol/l and don't show a refusal after information.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-05-26 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
one month survival | 1 month
  Survival at 1 month after the blood sample at the ED

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besançon, Besançon, France